CLINICAL TRIAL: NCT03627520
Title: Single-center, Open and Single-dose Clinical Trial to Explore the Mass Balance of Oral Suspension of 300 mg /100 μCi [14C] Sulfatinib in Chinese Adult Male Healthy Volunteers
Brief Title: A Mass Balance Study to Investigate the Absorption, Metabolism, and Excretion of [14C]Sulfatinib
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-012-00CH1
Record Dates: First submitted 2018-03-13; First posted 2018-08-13 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Intervention Model Description: This is single centre, open label, single dose study
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]Sulfatinib (Other): This is a single center and single dose in 6 volunteers. Subject would take a suspension containing 300 mg of Sulfatinib (containing about 100 μCi of radioactivity) within 1 hour after standard breakfast.
  Interventions: Drug: [14C]Sulfatinib

INTERVENTIONS:
Drug: [14C]Sulfatinib — 300 mg Sulfatinib with 100 µCi [14C]
  Other Names: 300 mg /100 μCi [14C] Sulfatinib, Sulfatinib, HMPL-012, Surufatinib

SUMMARY:
This is a single-center, open label and single-dose clinical trail, to explore the body mass balance and identify the major metabolites in Chinese adult male healthy volunteers after a single oral dose of [14C]Sulfatinib, to obtain the pharmacokinetic parameters of plasma and observe the safety of healthy volunteers after a single oral dose of [14C]Sulfatinib.

DETAILED DESCRIPTION:
In order to determine the optimal time point for sample collection, this study will be divided into two stages: the first stage, two volunteers will be enrolled, the volunteers should stop collecting the corresponding samples by the investigators based on radioactive test results, safety results combined with the actual comprehensive situation. And in the second stage sample collection time for another four volunteers will be determined and adjusted according to the results of the first stage.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF)
2. Age of 18-50 (inclusive)；
3. Body weight over 50 kg and body mass index (BMI) between 19-26 kg / m2 (inclusive)；

Exclusion Criteria:

1. Laboratory tests (blood tests, blood biochemical tests [fasting], coagulation tests, thyroid function tests, urinalysis, fecal occult blood) judged as clinically significant abnormal by investigators；
2. Clinically significant abnormal ECG at screening and before screening；
3. Hepatitis B surface antigen (HBsAg), e antigen (HBeAg) or hepatitis C antibody (HCV Ab) test positive；
4. Human immunodeficiency virus (HIV) antibody positive；
5. Treponema pallidum antibody positive.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Age of 18-50 (inclusive), Male
Enrollment: 6 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
To investigate the area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) of total radioactivity of [14C] Sulfatinib | Measured from the 0 hour to 216 hours
  The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration.

SECONDARY OUTCOMES:
To investigate the Maximum observed plasma concentration (Cmax) of total radioactivity of [14C] Sulfatinib | Measured from the 0 hour to 216 hours
  Maximum observed concentration, occurring at Tmax.
To investigate the time to Cmax (peak time, Tmax) of total radioactivity of [14C] Sulfatinib | Measured from the 0 hour to 216 hours
  The time at which maximum plasma concentration (Cmax) is observed.
To investigate Half-life (t1/2) of total radioactivity of [14C] Sulfatinib | Measured from the 0 hour to 216 hours
  The time at which Half-life (t1/2) is observed.
To obtain mass balance data after a single oral dose of [14C] Sulfatinib | Measured on the Day1 to Day15
  Quantitative analysis of total radioactivity in the excretion of Sulfatinib
To observe the safety of healthy volunteers after a single oral dose of [14C]Sulfatinib. | Measured from the date signed ICF to within 15 days after the single dose
  Adverse Event (AE) monitoring of [14C] Sulfatinib

CONTACTS AND LOCATIONS:
Overall Officials: Ke LI, PhD, Study Director — Hutchison Medipharma Ltd.
Locations (1):
- Hutchison Medipharma Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No